CLINICAL TRIAL: NCT05018533
Title: The Safety and Pharmacokinetics Study of TAKC-02 Inhalation Solution in Healthy Adult Males.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: TAK-Circulator Co. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TAKC-02-001
Record Dates: First submitted 2021-08-17; First posted 2021-08-24 (Actual); Last update posted 2022-06-02 (Actual); Status verified 2022-05

CONDITIONS: Healthy Volunteer
Keywords: antisense oligonucleotides; anti asthmatic agents

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Not applicable to a drug allotment and a dispensing staff
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (14):
- Cohort 1 (Experimental): TAKC-02 0.15mg Single dose
  Interventions: Drug: TAKC-02
- Placebo (to Cohort 1) (Placebo Comparator)
  Interventions: Drug: Placebo
- Cohort 2 (Experimental): TAKC-02 0.5mg Single dose
  Interventions: Drug: TAKC-02
- Placebo (to Cohort 2) (Placebo Comparator)
  Interventions: Drug: Placebo
- Cohort 3 (Experimental): TAKC-02 1.5mg Single dose
  Interventions: Drug: TAKC-02
- Placebo (to Cohort 3) (Placebo Comparator)
  Interventions: Drug: Placebo
- Cohort 4 (Experimental): TAKC-02 5mg Single dose
  Interventions: Drug: TAKC-02
- Placebo (to Cohort 4) (Placebo Comparator)
  Interventions: Drug: Placebo
- Cohort 5 (Experimental): TAKC-02 15mg Single dose
  Interventions: Drug: TAKC-02
- Placebo (to Cohort 5) (Placebo Comparator)
  Interventions: Drug: Placebo
- Cohort 6 (Experimental): TAKC-02 Multiple dose (low)
  Interventions: Drug: TAKC-02
- Placebo (to Cohort 6) (Placebo Comparator)
  Interventions: Drug: Placebo
- Cohort 7 (Experimental): TAKC-02 Multiple dose (high)
  Interventions: Drug: TAKC-02
- Placebo (to Cohort 7) (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TAKC-02 — Inhalation Solution
  Arms: Cohort 1; Cohort 2; Cohort 3; Cohort 4; Cohort 5; Cohort 6; Cohort 7
Drug: Placebo — Inhalation Solution
  Arms: Placebo (to Cohort 1); Placebo (to Cohort 2); Placebo (to Cohort 3); Placebo (to Cohort 4); Placebo (to Cohort 5); Placebo (to Cohort 6); Placebo (to Cohort 7)

SUMMARY:
MEX3B is an RNA-binding protein that is conserved in many animal species and has wide range of biological function. The MEX3B protein is deeply involved in the expression of various cytokines associated with the onset and exacerbation of several diseases such as inflammatory diseases, metabolic diseases, and malignant tumors. TAKC-02 is a nucleic acid medicine, antisense oligonucleotide, inhibits the MEX3B synthesis expected to have potential as new medication.

This plans to evaluate the safety profile of the inhalation solution in order to develop TAKC-02 for severe asthma.

The study is a double-blind, randomized, placebo-controlled Phase I study. The primary objective of the study is to assess the safety and tolerability of single and multiple inhaled doses of TAKC-02 in healthy male subjects. The study is a Single Ascending Dose (Step 1) followed by a Multiple Comparative Dose (Step 2).

DETAILED DESCRIPTION:
This initial Phase I study will be conducted in normal healthy male volunteers to obtain an unconfounded understanding of the safety, tolerability and pharmacokinetics of TAKC-02 inhalation solution. TAKC-02 is being developed as a medication for uncontrolled severe asthma. The first-in-human, randomized, double-blind trial will evaluate single ascending doses (SAD) and subsequently multiple ascending doses (MAD) of TAKC-02 and placebo.

Step 1 (SAD) :

There will be 5 cohort of 6 (Cohort 1, 2, 3) or 8 (Cohort 4, 5) subjects each. Subjects in each cohort are randomized in a 2:1 ratio (Cohort 1, 2, 3) and 3:1 ratio to receive a single dose of the study drugs, TAKC-02 or Placebo. The SAD study will evaluate the safety and tolerability of a single dose of TAKC-02 and determine the starting and maximum doses for Step 2. Pharmacokinetics will be also analyzed. One cohort (cohort 4.5) maybe added depending on the incidence of adverse effect in the lower dosing group.

Step 2 There will be 2 cohort f 8 subjects each. Subjects in both cohorts are randomized in a 3:1 ratio to receive multiple doses of the study drugs, TAKC-02 or Placebo. The safety and tolerability of repeated administration of TAKC-02 for 2 weeks will be evaluated, and the maximum dose of this drug in the next phase will be estimated. Pharmacokinetics will be also analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Both Step 1 and Step 2 are for healthy adult males who meet all of the following conditions.

  1. Subjects are normal healthy men
  2. Aged between 20 and 40 at the time of consent
  3. Subjects who have obtained the voluntary consent of the person in writing
  4. Subjects with BMI of 18.5 or more and less than 25.0 kg / m2
  5. Subjects who can be hospitalized during the cohort transition safety assessment period

Exclusion Criteria:

* Both Step 1 and Step 2 do not apply to those who meet any of the following conditions.

  1. Subjects with clinically problematic complications or medical history
  2. Subjects with a history of drug allergies
  3. Smokers (those who have smoked within 1 year)
  4. Subjects with hypersensitivity disease (excluding asymptomatic pollinosis)
  5. Those who may affect the absorption, distribution, metabolism and excretion of drugs
  6. Subjects have been prescribed a drug intended for treatment within 4 weeks before administration of the study drug, or those who need administration during the period of participation in the study
  7. Subjects have used over-the-counter drugs within 4 weeks before administration of the study drug, or those who need to use it during the period of participation in the study
  8. Subjects ingested alcoholic beverages or caffeine-containing beverages within 24 hours before administration of the study drug
  9. Subjects with reduced lung function (FEV1.0% <70%)
  10. Subjects with alcoholism or drug addiction
  11. Subjects have a positive reaction in the substance abuse test
  12. Subjects tested positive for HBsAg, hepatitis C virus (HCV) antibody, HIV antigen / antibody, syphilis serum reaction or severe acute respiratory syndrome (SARS)-CoV-2 nucleic acid amplification
  13. Subjects collected 400 mL or more of whole blood within 16 weeks before administration of the study drug or 200 mL or more of blood within 4 weeks, or those who collected component blood (plasma component and platelet component) within 2 weeks before administration of the study drug, or subjects whose annual total blood collection volume exceeds 1200 mL, including the planned blood collection volume for clinical trials
  14. Subjects have been treated with TAKC-02 in the past
  15. Subjects participated in another clinical trial and were administered anther test drug within 16 weeks before the administration of the study drug, or those who participated in another clinical trial at the same time as this clinical trial.
  16. Subjects have been vaccinated against new coronavirus, influenza, etc. within 4 weeks before the administration of the study drug, or who are scheduled to be vaccinated during the period of participation in the study.
  17. Subjects are not willing to adhere to proper contraception using effective contraception for 3 weeks after the last dose of the study drug from the date of admission of study site.
  18. Subjects are judged inappropriate to participate in the clinical trial by the investigator or the co-investigator.

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2021-08-17 (Actual); Primary Completion 2021-12-28 (Actual); Study Completion 2021-12-28 (Actual)

PRIMARY OUTCOMES:
Changes in the rate of adverse events | Up to 7 days after dose
  assessed by the change in number of adverse events

SECONDARY OUTCOMES:
AUC from time zero to the time of the last quantifiable concentration (AUC0-t last) | Up to 48 hours after last dose
Cmax | Up to 48 hours after last dose
Tmax | Up to 48 hours after last dose
T1/2 | Up to 48 hours after last dose

CONTACTS AND LOCATIONS:
Locations (1):
- TAKC-02 Study Site, Tokyo, Japan